CLINICAL TRIAL: NCT02786693
Title: Evaluation of Diagnosis of Fever and Biologic Inflammatory Syndrome of Unknown Origin
Acronym: FUO
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A01627-42
Record Dates: First submitted 2016-01-08; First posted 2016-06-01 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Fever of Unknown Origin
Keywords: TEP-scan
MeSH Terms: conditions — Fever of Unknown Origin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FUO and SII patients: Patients with fever > 38,3°C for more than a week, OR CRP> 5mg/L, without diagnosis after a first step clinical examination and paraclinical exams.

SUMMARY:
Fever of unknown origin (FUO) and biologic inflammatory syndrome of unknown origin (SII) are two frequent causes of hospitalization or consultation in infectious disease unit and internal medicine.

There are many etiologies, in four categories: infections, auto-immune disease, cancer and miscellaneous causes. Currently there is no specifics recommendations to follow a "diagnosis way" of FUO and SII.

Purpose: Evaluation of clinical practices in the diagnosis of fever and biologic inflammatory syndrome of unknown origin, in two units of the University Grenoble Hospital.

DETAILED DESCRIPTION:
Fever of unknown origin (FUO) and biologic inflammatory syndrome of unknown origin (SII) are two frequent causes of hospitalization or consultation in infectious disease unit and internal medicine unit.

The initial definition for FUO was proposed by Petersdorf and Beeson in 1961 : "fever > 38,3°C, permanent or recurrent, for more than 3 weeks, without diagnosis after one week hospitalisation and explorations". This definition has been updated by Durack and Street in 1991 who distinguish "classics FUO" from 3 other categories : nosocomial, patient with HIV and neutropenia. They also choose an other way of diagnosis : 3 days of investigations in hospital OR in consultation.

Finally, Knokaert and al. proposed a new definition, based on a qualitative criterion: No diagnosis after a first step and complete clinical and paraclinical check up.

The evolution of FUO's prevalence is not describe so much. There are many etiologies, classified in four categories: infections, auto-immune disease, cancer and miscellaneous causes. The distribution of FUO's causes may change according to geographical localisation, and seems to evolve over time, with apparition of new infectious and inflammatory diseases, and the advent of new diagnosis tools.

Currently there is no specifics recommendations to follow a "diagnosis way" of FUO and SII. It starts with a complete physical examination and some first lign further exams. Without diagnosis, paraclinical explorations are continued with more specific exams, according to the presence or the absence of diagnosis clues.

The TEP scanner has shown a great value in the diagnosis of FUO, and trend to be more performed.

Investigators propose to evaluate professional practices in the diagnosis of fever and biologic inflammatory syndrome of unknown origin, and especially the interest of TEP Scan, in two units of the University Grenoble Hospital.

Investigators will study prevalence of FUO and SII, and of each causes of FUO and SII, and the prognosis of patients with FUO and SII, according to the presence or the absence of final diagnosis, as well as the economic impact of the different complementary exams.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old
* with fever> 38.5°C and/or CRP> 5mg/L for more than a week
* with standard check-up that did not allow a causal diagnosis

Exclusion Criteria:

* immunosuppression : HIV, neutropenia, known cancer with chemotherapy, immunosuppressive treatment or corticotherapy (> 10mg/L for >3 weeks)
* nosocomial fever
* pregnant women
* patients who are not able to sign a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with fever and biologic inflammatory syndrome of unknown origin for more than a week
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Presence of a final diagnosis after paraclinical explorations | 1 year
  Final diagnosis according to the previous classification : infectious disease, inflammatory or auto-immune disease, cancer, or miscellaneous cause.

SECONDARY OUTCOMES:
prevalence of FUO/SII : | 1 year
  Number of patients with FUO and SII, assessed by inclusion in the present study .
causes of FUO/SII: Proportion of each causes of FUO/SII, according to the main outcome after final diagnosis | 1 year
  5 possible causes : infectious diseases, auto-immune and inflammatory diseases, cancers, miscellaneous causes.
  Final diagnosis is determined according to the usual criteria, reviewed by two practitioners.
Mortality rate of patient with FUO and SII, according to the presence or absence of a final diagnosis | 1 year
  mortality rate
Medical economic evaluation of the utility of the TEP scan in the diagnostic approach | 1 year
  Benefit of TEP Scan in the diagnosis of FUO and SII : The utility is defined as an examination which allows :
  * the direct diagnosis or
  * direct the examination which will allow the diagnosis. The utility will be validated for every examination by 2 responsible doctors

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Bouillet, PhD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - CHU Grenoble, Grenoble
  - University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] PETERSDORF RG, BEESON PB. Fever of unexplained origin: report on 100 cases. Medicine (Baltimore). 1961 Feb;40:1-30. doi: 10.1097/00005792-196102000-00001. No abstract available. PMID 13734791
- [Background] Durack DT, Street AC. Fever of unknown origin--reexamined and redefined. Curr Clin Top Infect Dis. 1991;11:35-51. No abstract available. PMID 1651090
- [Background] Knockaert DC, Vanderschueren S, Blockmans D. Fever of unknown origin in adults: 40 years on. J Intern Med. 2003 Mar;253(3):263-75. doi: 10.1046/j.1365-2796.2003.01120.x. PMID 12603493
- [Background] Bleeker-Rovers CP, Vos FJ, de Kleijn EMHA, Mudde AH, Dofferhoff TSM, Richter C, Smilde TJ, Krabbe PFM, Oyen WJG, van der Meer JWM. A prospective multicenter study on fever of unknown origin: the yield of a structured diagnostic protocol. Medicine (Baltimore). 2007 Jan;86(1):26-38. doi: 10.1097/MD.0b013e31802fe858. PMID 17220753
- [Background] Kucukardali Y, Oncul O, Cavuslu S, Danaci M, Calangu S, Erdem H, Topcu AW, Adibelli Z, Akova M, Karaali EA, Ozel AM, Bolaman Z, Caka B, Cetin B, Coban E, Karabay O, Karakoc C, Karan MA, Korkmaz S, Sahin GO, Pahsa A, Sirmatel F, Solmazgul E, Ozmen N, Tokatli I, Uzun C, Yakupoglu G, Besirbellioglu BA, Gul HC; Fever of Unknown Origin Study Group. The spectrum of diseases causing fever of unknown origin in Turkey: a multicenter study. Int J Infect Dis. 2008 Jan;12(1):71-9. doi: 10.1016/j.ijid.2007.04.013. Epub 2007 Jul 12. PMID 17629532
- See also: university hospital Grenoble website — http://www.chu-grenoble.fr